CLINICAL TRIAL: NCT02589730
Title: Individualized Management Based on Mobile Phone Platform in Diabetic Patients
Brief Title: Effect of Smart Phone Application on the Individualized Management of Chinese Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Geping Information Technology Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IMME-6Y01
Record Dates: First submitted 2015-10-16; First posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus
Keywords: Smartphone app; diabetic management; lifestyle behaviors; medication management
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- online mutual management (Experimental): The patients received the online coaching of a doctor and diabetes educator via smart phone based welltang app.
  Interventions: Device: Welltang App
- online self-management (Experimental): The patients received the online coaching of a doctor alone via smart phone based welltang app.
  Interventions: Device: Welltang App
- hospital regular management (No Intervention): The patients received usual care and did not use smart phone.

INTERVENTIONS:
Device: Welltang App — This App is a large platform of individualized diabetic management
  Arms: online mutual management; online self-management

SUMMARY:
The purpose of this study was to explore a model suitable for the individualized diabetic management based on the mobile application coaching and demonstrate its effect among the diabetic mellitus population.

DETAILED DESCRIPTION:
The enrolled patients will be randomly divided into three groups: group of online self management, group of online mutual management and the control group. The estimated sample size was 78 patients for each group. All the patients attend two follow-up visits at the hospital, after 3 and 6 months. The data will be collected by a full-time recorder and analyzed using specific statistical software. The enumeration data are analyzed by chi-square test, while the measurement data are analyzed by one-way ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of DM for more than 6 months;
* Glycated hemoglobin more than or equal to 8% within 3 months;
* Age:18-65 years.

Exclusion Criteria:

* Insulin pump users;
* Pregnant;
* Active substance, alcohol, or drug abuser;
* Psychotic or schizophrenic under active care;
* Severe hearing or visual impairment and other complications;
* Drug users (such as glucocorticoid or thyroid hormone) 3 months before the enrollment;
* No smartphone access.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
change in glycated hemoglobin levels | six months

SECONDARY OUTCOMES:
change in lipid profile levels | six months
change of urinary albumin creatinine rate | six months
change of hepatic function | six months
change of blood creatine | six months
change of blood urea nitrogen | six months
change in scores measured by MKT | six months

OTHER OUTCOMES:
change in scores measured by SDSCA | six months
change in scores measured by DES-SF | six months
change in scores measured by Morisky | six months
change in scores measured by self distress scale | six months
change in scores measured by self anxiety scale | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Six People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang L, He X, Shen Y, Yu H, Pan J, Zhu W, Zhou J, Bao Y. Effectiveness of Smartphone App-Based Interactive Management on Glycemic Control in Chinese Patients With Poorly Controlled Diabetes: Randomized Controlled Trial. J Med Internet Res. 2019 Dec 9;21(12):e15401. doi: 10.2196/15401. PMID 31815677